CLINICAL TRIAL: NCT05025657
Title: Advocates for All Youth
Acronym: ALLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-3790
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Depression, Anxiety; Self Efficacy; Suicidal Ideation
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program (Experimental)
  Interventions: Behavioral: ALLY
- Control (Placebo Comparator)
  Interventions: Behavioral: ALLY

INTERVENTIONS:
Behavioral: ALLY — ALLY is a universal, school-based prevention program that takes place during the school day with individual students over 6 weeks.

SUMMARY:
Advocates for ALLY Youth (ALLY) is a universal, school-based, multicomponent positive psychology program aimed to increase youth's well-being and reduce symptoms of psychological distress including depression, anxiety, and stress.

ELIGIBILITY:
Inclusion Criteria:

* students enrolled at participating schools

Exclusion Criteria:

* none

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of Anxiety and Depression | 3 months
  The PROMIS Emotional Distress Anxiety and PROMIS Emotional Distress Depressive Symptoms scales (Irwin et al., 2010) were used to assess negative affectivity. Each 8-item short form elicits responses from the student on a 5-point Likert scale from "never" to "always" over the past 7-day period. The items are summed for a score ranging from 8 to 40 with higher scores indicating more elevated negative affectivity. Scores are then translated to T-scores, with T-scores below 55 classified as "normal," T-scores between 55 and 60 classified as "mild," T-scores between 60 and 70 classified as "moderate," and T-scores above 70 classified as "severe." The measure demonstrated satisfactory goodness of fit and adequate internal reliability (α = 0.85) in children and adolescents aged 8-17 years (Irwin et al., 2010). Elevated negative affectivity was endorsed in cases when students scored mild or higher for symptoms of both depression and anxiety on each of the PROMIS scales.

SECONDARY OUTCOMES:
Self-efficacy | 3 months
  The Self-Efficacy Questionnaire for Children (SEQ-C) validated among adolescents aged 12-19 years was used to assess self-efficacy (Muris, 2001). This 24-item survey assesses three key domains of self-efficacy: (1) social self-efficacy, defined as perceived capability for peer relationships and assertiveness; (2) academic self-efficacy, which is the perceived capability to manage one's own learning behavior, to master academic subjects, and to fulfill academic expectations; and (3) emotional self-efficacy, which is the perceived capability of coping with negative emotions. Each item is scored on a 5-point Likert scale ranging from "not at all" to "very well." Subscale scores and an overall or total self-efficacy score are obtained by summing respective items, with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Loachapoka Elementary School, Loachapoka, Alabama, United States

IPD SHARING:
Plan to Share IPD: No